CLINICAL TRIAL: NCT00176930
Title: Allogeneic Transplant for Hematological Malignancy
Brief Title: Stem Cell Transplant for Hematological Malignancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: replaced by another study ; Trial re-written as MT2015-29
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001LS049; MT2001-02 (Other: Blood and Marrow Transplantation Program); 0107M05202 (Other: IRB, University of Minnesota); NCT00393133 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Leukemia, Myeloid, Chronic; AML; Leukemia, Lymphocytic, Acute; MDS; Leukemia, Lymphocytic, Chronic; JMML; Hodgkin's Disease; Non-hodgkin's Lymphoma; Multiple Myeloma
Keywords: stem cell transplant; chronic leukemia; acute leukemia; irradiation; chemotherapy
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Cyclophosphamide; Whole-Body Irradiation; Radiotherapy; Busulfan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- PBSC: No TBI (Experimental): Patients who are not able to receive Total Body Irradiation (TBI) receives cyclophosphamide, Busulfan and Peripheral Blood Stem Cells (PBSC) as a source of transplant
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Drug: Busulfan
- Marrow : No TBI (Experimental): Patients who are not able to receive Total Body Irradiation (TBI) receives cyclophosphamide, Busulfan and Bone Marrow as a source of stem cell transplant
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Drug: Busulfan
- UCB : No TBI (Experimental): Patients who are not able to receive Total Body Irradiation (TBI) receives cyclophosphamide, Busulfan and Umbilical Cord Blood (UCB) as a source of stem cell transplant
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Drug: Busulfan
- UCB : No TBI/Bu/Cy/ATG (Experimental): Patients who receives Umbilical Cord Blood (UCB) as a source of transplant and who have not had chemotherapy in the prior 3 months receives ATG in addition to cyclophosphamide, Busulfan preparative regimen
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Drug: Busulfan; Drug: Equine ATG (ATGAM)
- PBSC (Experimental): Patients receiving cyclophosphamide, Total Body Irradiation (TBI) and Peripheral blood stem cells as a source of transplant
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Radiation: Total Body Irradiation
- Marrow (Experimental): Patients receiving cyclophosphamide, Total Body Irradiation (TBI) and Bone Marrow as a source of stem cell transplant
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Radiation: Total Body Irradiation
- UCB (Experimental): Patients receiving cyclophosphamide, Total Body Irradiation (TBI), and Umbilical Cord Blood (UCB) as a source of stem cell transplant
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Radiation: Total Body Irradiation
- Co-Enroll From MT0403 (Experimental): Patients receiving cyclophosphamide, Total Body Irradiation (TBI) , CD4+CD25+ and Peripheral Blood Stem Cells (PBSC) as a source of transplant. These patients are co-enrolled on the MT2004-03 trial (NCT00725062)
  Interventions: Biological: Stem Cell Transplant; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Biological: CD4+/CD25+ cells

INTERVENTIONS:
Biological: Stem Cell Transplant — Certain cancers can be treated by giving patients stem cells that come from someone else. This is called a stem-cell transplant. As part of the transplant process, patients receive high doses of chemotherapy and/or radiation to treat their underlying disease, such as cancer. As one of its effects, this treatment also kills the healthy stem cells that are already in the marrow. The transplant provides new stem cells for the patient from a healthy donor; that replace the bone marrow and allow the blood counts to recover. (Allowable sources of stem cells = related or unrelated bone marrow or peripheral blood, for Busulfan/cyclophosphamide/ATG preparative chemo only, umbilical cord blood is also permitted.)
  Other Names: Bone Marrow Transplant.
Drug: Cyclophosphamide — 60 mg/kg intravenously (IV) Days -6 and -5 or 50 mg/kg/day IV Days -5 through -2.
  Other Names: Cytoxan
Radiation: Total Body Irradiation — On Day -4, -3, -2, -1 total body irradiation is given twice daily.
  Other Names: Radiation therapy
  Arms: Co-Enroll From MT0403; Marrow; PBSC; UCB
Drug: Busulfan — When not receiving total body irradiation, administered Days -9 through -6, 0.8 mg/kg/dose by intravenous dosing every 6 hours.
  Other Names: Busulfex; Myleran
  Arms: Marrow : No TBI; PBSC: No TBI; UCB : No TBI; UCB : No TBI/Bu/Cy/ATG
Drug: Equine ATG (ATGAM) — UCB recipients who have not had chemotherapy in the preceding 3 months will also receive Equine ATG (ATGAM) 15 mg/kg IV will be administered every 12 hours for 6 doses beginning on day -3 per institutional guidelines
  Arms: UCB : No TBI/Bu/Cy/ATG
Biological: CD4+/CD25+ cells — On days -2, patients will receive CD4+/CD25+ cells intravenously.
  Arms: Co-Enroll From MT0403

SUMMARY:
The purpose of this study is to develop a standard of care treatment using allogeneic stem cells for patients with cancers of the blood.

The protocol was revised to reflect that this study is considered "treatment guidelines", rather than a research study.

DETAILED DESCRIPTION:
Preparative regimen using total body irradiation (TBI) and cyclophosphamide:

1. on day -6 and -5: cyclophosphamide is given,
2. on day -4, -3, -2, and -1: TBI is given,
3. on day 0: stem cell or bone marrow is infused.

Alternate preparative therapy for patients not able to receive TBI

The chemotherapy (cyclophosphamide and busulfan) is given with the intent of destroying the bone marrow, eliminating any cancerous and preparing for the transplant of the donor's blood stem cells by suppressing the immune system.

l. Ten days before the transplant (Day 10), subjects will be admitted to the bone marrow transplant unit and placed in isolation to reduce exposure to infections. Isolation will be continued until adequate numbers of cells are present in the blood to fight infection.

2. On day -9, -8, -7, -6 busulfan is given.

3. On day -5, -4, -3, -2 cyclophosphamide is given.

4. On day -1 no therapy is given (day of rest).

5. On day 0 the donor stem cells are given intravenously. Additional cells may be given on day +1 or 2 as needed.

Transplant:

Subjects will be admitted to the bone marrow transplant unit and put in isolation to reduce exposure to infectious agents. During this time, they will receive the preparative treatment outlined above. Once they have received the preparative regimen, stem cells will be obtained from the donor and given intravenously.

The new stem cells will replace the bone marrow that was damaged by the treatment for the cancer.

Isolation will be continued until adequate numbers of cells are present in the blood to fight infection. Subjects will then be transferred from the bone marrow transplant unit and discharged from the hospital when medically ready. Subjects will be expected to return for follow-up to the bone marrow transplant clinic at specific dates as determined by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Donor will be <75 years of age and in good health.
* Recipients will be < or = 55 years, will have normal organ function (excluding bone marrow) and will have a Karnofsky activity assessment > or = 90%.
* Recipients with related or unrelated donor matched at the HLA A, B, DRB1 loci, or mismatched related or unrelated (if < 35 years old) at a single HLA A, B, DRB1 locus.
* Recipients will be eligible in one of the following disease categories
* Chronic myelogenous leukemia in accelerated phase or in post blast crisis second or greater chronic phase; or in chronic phase but intolerant of or resistant to tyrosine kinase inhibitors.
* Acute myelocytic leukemia in first or greater remission, or first, second or third relapse.
* Acute lymphocytic leukemia in the 2nd or greater bone marrow remission.
* High risk children will be transplanted in first remission if they meet criteria
* Myelodysplastic syndrome.
* Myeloproliferative Diseases - (i.e. myelofibrosis, chronic myelomonocytic leukemia (CMML))
* Juvenile myelomonocytic leukemia
* Chronic lymphocytic leukemia
* Advanced non-Hodgkin's (NHL).
* Advanced Hodgkin's disease beyond PR2 (> CR3, > PR3).
* Multiple Myeloma after initial therapy.
* Donors and recipients signed informed consent

Exclusion Criteria

donors and recipients should meet the following test criteria.

* required for donors:

  * anti-HIV, Hepatitis B, surface antigen, anti-HCV, CMV, HSV, EBV serologies, pre-priming.
  * CBC, platelet count each day of apheresis, day 0 (or 1 or 2 as needed)
* required for recipients:

  * anti-HIV, Hepatitis B, surface antigen, anti-HCV, CMV, HSV, EBV serologies, pre-transplant.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 330 (Actual)
Dates: Start 2001-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weisdorf, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient withdrew consent.
Groups:
- Umbilical Cord Blood: Patients receiving cyclophosphamide, Total Body Irradiation (TBI), and Umbilical Cord Blood (UCB) as a source of stem cell transplant
  Cyclophosphamide: 60 mg/kg intravenously (IV) Days -6 and -5 or 50 mg/kg/day IV Days -5 through -2.
  Total Body Irradiation: On Day -4, -3, -2, -1 total body irradiation is given twice daily.
- Co-Enroll From MT0403: Patients receiving cyclophosphamide, Total Body Irradiation (TBI) , CD4+CD25+ and Peripheral Blood Stem Cells (PBSC) as a source of transplant. These patients are co-enrolled on the MT2004-03 trial (NCT00725062)
  Cyclophosphamide: 60 mg/kg intravenously (IV) Days -6 and -5 or 50 mg/kg/day IV Days -5 through -2.
  Total Body Irradiation: On Day -4, -3, -2, -1 total body irradiation is given twice daily. CD4+/CD25+ cells: On days -2, patients will receive CD4+/CD25+ cells intravenously.
Period: Overall Study
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Started | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Completed | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Umbilical Cord Blood: Patients receiving cyclophosphamide, Total Body Irradiation (TBI), and Umbilical Cord Blood (UCB) as a source of stem cell transplant
- Total: Total of all reporting groups
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403 | Total
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2 | 329
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 12 | 0 | 0 | 9 | 51 | 2 | 2 | 76
  Between 18 and 65 years | 12 | 1 | 1 | 1 | 204 | 34 | 0 | 0 | 253
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 0 | 1 | 78 | 35 | 1 | 1 | 130
  Male | 2 | 9 | 1 | 0 | 135 | 50 | 1 | 1 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 5
  Not Hispanic or Latino | 5 | 11 | 1 | 1 | 82 | 41 | 2 | 2 | 145
  Unknown or Not Reported | 7 | 2 | 0 | 0 | 130 | 40 | 0 | 0 | 179
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 7
  Asian | 0 | 0 | 0 | 0 | 6 | 4 | 0 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 5 | 3 | 0 | 0 | 8
  White | 11 | 13 | 1 | 1 | 178 | 64 | 2 | 2 | 272
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 20 | 10 | 0 | 0 | 31
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2 | 329

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Disease-Free Survival at 2 Years Post Transplant
Description: Disease-Free Survival is the length of time during and after medication or treatment during which the disease being treated (usually cancer) does not get worse. It is sometimes used as a metric to study the health of a person with a disease to try to determine how well a new treatment is working.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 4 | 9 | 0 | 0 | 100 | 52 | 2 | 2

2. Primary Outcome: Number of Participants Experiencing Disease-Free Survival at 5 Years Post Transplant
Description: as for outcome 1
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 3 | 9 | 0 | 0 | 85 | 48 | 2 | 2

3. Secondary Outcome: Number of Participants With Neutrophil Engraftment
Description: Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm^3 (0.5 x 10^9/L) or greater.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 11 | 13 | 0 | 1 | 206 | 83 | 2 | 2

4. Secondary Outcome: Number of Participants With Acute Graft-versus-host Disease (GVHD)
Description: Acute Graft-Versus-Host Disease (aGVHD) is a severe short-term complication created by infusion of donor cells into a foreign host. Determine the incidence of grade II-IV acute graft-versus-host disease (GVHD) at day 100 post transplant. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria used for staging.
  Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 6 | 2 | 1 | 0 | 89 | 23 | 0 | 0

5. Secondary Outcome: Number of Participants With Chronic Graft-Versus-Host Disease
Description: Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host. Determine the incidence of chronic GVHD 1 year post transplant. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria. Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 4 | 2 | 0 | 0 | 87 | 14 | 0 | 1

6. Secondary Outcome: Number of Participants With Persistence or Relapse of Malignancy at 2 Years Post Transplant
Description: Defined as the return of disease after its apparent recovery/cessation. Patients with leukemia and lymphoma involving the BM and multiple myeloma will have this done by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients with lymphoma and myeloma will have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 3 | 4 | 0 | 0 | 63 | 17 | 0 | 0

7. Secondary Outcome: Number of Participants With Persistence or Relapse of Malignancy at 5 Years Post Transplant
Description: as for outcome 6
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 4 | 4 | 0 | 0 | 69 | 20 | 0 | 0

8. Secondary Outcome: Number of Participants Who Were Alive at 2 Year Post Transplant
Description: The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 5 | 11 | 0 | 0 | 122 | 59 | 2 | 2

9. Secondary Outcome: Number of Participants Who Were Alive at 5 Year Post Transplant
Description: as for outcome 8
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 3 | 9 | 0 | 0 | 100 | 54 | 2 | 2

10. Secondary Outcome: Number of Participants Experiencing Engraftment Failure
Description: Graft failure is defined as not accepting donated cells. The donated cells do not make the new white blood cells, red blood cells and platelets.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
Number analyzed (Participants) | 12 | 13 | 1 | 1 | 213 | 85 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | PBSC: No TBI | Marrow : No TBI | UCB : No TBI | UCB : No TBI/Bu/Cy/ATG | PBSC | Marrow | Umbilical Cord Blood | Co-Enroll From MT0403
All-Cause Mortality (participants affected / at risk) | 9/12 | 4/13 | 1/1 | 1/1 | 113/213 | 31/85 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/13 | 0/1 | 0/1 | 32/213 | 10/85 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 12/12 | 10/13 | 1/1 | 1/1 | 183/213 | 71/85 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBSC: No TBI (N=12) | Marrow : No TBI (N=13) | UCB : No TBI (N=1) | UCB : No TBI/Bu/Cy/ATG (N=1) | PBSC (N=213) | Marrow (N=85) | Umbilical Cord Blood (N=2) | Co-Enroll From MT0403 (N=2)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Primary Graft Failure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 20 (20) | 8 (8) | 0 (0) | 0 (0)
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 0 (0) | 0 (0)
Syndromes (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Death due to accident (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBSC: No TBI (N=12) | Marrow : No TBI (N=13) | UCB : No TBI (N=1) | UCB : No TBI/Bu/Cy/ATG (N=1) | PBSC (N=213) | Marrow (N=85) | Umbilical Cord Blood (N=2) | Co-Enroll From MT0403 (N=2)
Infection (Infections and infestations) | 10 (37) | 9 (32) | 1 (6) | 1 (4) | 114 (375) | 54 (169) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (14) | 6 (8) | 1 (14) | 1 (1) | 91 (143) | 42 (70) | 1 (1) | 2 (7)
Intubation (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 34 (45) | 14 (22) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 26 (27) | 21 (23) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 25 (25) | 11 (11) | 0 (0) | 0 (0)
Elevated Liver Function Tests (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 25 (26) | 10 (11) | 0 (0) | 0 (0)
GI Bleeding (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 24 (26) | 6 (7) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 12 (12) | 13 (13) | 0 (0) | 1 (2)
Dialysis (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 16 (16) | 8 (12) | 0 (0) | 0 (0)
Veno occlusive disease (VOD) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 15 (18) | 7 (10) | 0 (0) | 0 (0)
Pumonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 16 (18) | 7 (7) | 0 (0) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 16 (16) | 7 (8) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 14 (15) | 5 (5) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 8 (8) | 6 (7) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 3 (3) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 13 (13) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 4 (4) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 6 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT00176930/Prot_SAP_000.pdf